# Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines – Montelukast vs Fluticasone

NCT05457855

July 10, 2023

## 1. Comparison Details

## a. Intended aim(s)

To evaluate the comparative risk of dementia onset between patients treated with <u>Montelukast versus Fluticasone</u> for asthma.

## b. Primary endpoint

Incident dementia (i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere).

## 2. Person responsible for implementation

Seanna Vine

## 3. Data Source(s)

Medicare, 2008-2018

## 4. Study Design Diagrams





### 5. Cohort Identification

## a. Cohort Summary

This study will employ a new user, active comparator, observational cohort study design comparing <u>Montelukast versus Fluticasone</u>. The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of study drugs (cohort entry/index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).

## b. Key details regarding cohort creation

### Index date:

• Day of initiation of new Montelukast versus Fluticasone use

## Inclusion criteria for analyses 1, 3, 4:

- Aged > 65 years on the index date
- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage
- No use of <u>Montelukast versus Fluticasone</u>, any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date
- No history of nursing home admission recorded in any time prior to and including index date
- At least two claims with asthma diagnosis recorded in 365 days prior to index date (ICD-9 493.0x, 493.1, 493.2x, 493.8x, 493.9x or ICD-10 J44.0, J44.1, J44.9, J45.2x, J45.3x, J45.4x, J45.5x, J45.9x)

## Inclusion criteria for analysis 2:

- Aged > 65 years on the index date
- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage or 365 days registration with a practice contributing data to CPRD prior to index date
- No use of <u>Montelukast versus Fluticasone</u>, any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date
- No history of nursing home admission recorded in any time prior to and including index date
- At least two claims with asthma diagnosis recorded in 365 days prior to index date (ICD-9 493.0x, 493.1,

493.2x, 493.8x, 493.9x or ICD-10 J44.0, J44.1, J44.9, J45.2x, J45.3x, J45.4x, J45.5x, J45.9x)

• 180-day continuous use of Montelukast versus Fluticasone starting on the index date

# c. Flowchart of the study cohort assembly

| | Less Excluded Patients | Remaining Patients |
|---|---|---|
| All patients | | 23,466,175 |
| Did not meet cohort entry criteria | -21,749,739 | 1,716,436 |
| Excluded due to insufficient enrollment | -1,010,844 | 705,592 |
| Excluded based on Dementia Exclusion | -113,159 | 592,433 |
| Excluded based on Nursing Home Admission | -62,588 | 529,845 |
| Excluded based on Peripheral artery disease Diagnosis | -454,167 | 75,678 |
| Excluded anyone aged <65 at index | -24,145 | 51,533 |
| Patients in Montelukast group | | 12,575 |
| Patients in Fluticasone group | | 38,958 |
| Final cohort | | 51,533 |

# 6. Variables

# a. Exposure-related variables:

Study drug:

The study exposure of interest is initiation of Montelukast

Comparator: Fluticasone

# b. Covariates:

| Demographics | |
|--------------|-----------------------------|
| Age | Region |
| Gender | Calendar year of index date |
| Race | Low income subsidy |

| Dementia risk factors | |
|-------------------------|------------------|
| Diabetes Depression | |
| Obesity | Anxiety |
| Hypertension | Bipolar disorder |
| Coronary artery disease | Schizophrenia |

| Markers for healthy behavior, frailty, healthcare use | |
|---|---|
| Smoking Number of outpatient visits | |
| Mammography | Number of hospitalizations |
| Colonoscopy Number of serum creatinine tests ordered | |
| Fecal occult blood test | Composite frailty score |
| Influenza vaccination Number of C-reactive protein tests | |
| Pneumococcal vaccination | Osteoporosis |
| Herpes zoster vaccination | Fractures |
| Bone mineral density test | Falls |

| Number of distinct generic agents | Use of supplemental oxygen |
|-----------------------------------|----------------------------|
| Number of emergency room visits | Combined comorbidity score |

| Other Asthma treatments and Asthma severity indicators | |
|---|---|
| Respiratory failure | LABA |
| Asthma exacerbation | SABA |
| Tuberculosis | SAMA |
| Lung Cancer | LAMA |
| Bronchiectasis | ICS (excluding Fluticasone) |
| Sarcoidosis | Omalizumab, Mepolizumab, Reslizumab, |
| | Benralizumab, Dupilumab |
| Pulmonary Hypertension | Leukotriene receptor antagonist (excluding |
| | Montelukast) |
| Interstitial lung disease, lung fibrosis, ARDS | Number of Pulmonologist visits |
| Acute Upper/ Lower Respiratory Tract infection | Pulmonary function test |
| Pneumonia | Antibiotics |
| Corticosteroids | |

| Comedication use | |
|---|---|
| Lithium | Diuretics |
| Anti-epileptic mood stabilizers | Nitrates |
| Anti-epileptics (other than mood stabilizers) | Lipid lowering drugs |
| Atypical antipsychotics | Non-insulin diabetes medications |
| Benzodiazepines | Insulin |
| Serotonin-norepinephrine reuptake Inhibitors | Antidepressants |
| Selective serotonin reuptake inhibitors | Angiotensin II receptor blockers (ARBs) |
| Tricyclic antidepressants (TCAs) | Angiotensin converting enzyme inhibitors (ACEi) |
| Typical antipsychotics | Calcium channel blockers |
| Anticoagulants | Beta blockers |
| Antiplatelet agents | Disease-modifying antirheumatic drugs (DMARDs) |

| Comorbid conditions | |
|---|---|
| Atrial fibrillation | Ischemic heart disease |
| Coronary artery disease | Chronic obstructive pulmonary disease |
| Heart failure | Malignancy |
| Stroke or transient ischemic attack | Drug or alcohol abuse or dependence |
| Peripheral vascular disease | Venous thromboembolism |
| Hyperlipidemia | Chronic liver disease |
| Renal dysfunction Rheumatoid Arthritis | |

ICD-9, ICD-10, HCPCS, and NDC codes used to define the covariates listed above are available in Appendix A.

- c. Outcome variables and study follow-up:
- <u>Primary outcome</u>: incident dementia, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Outcome will be defined by 1 inpatient claim or 2 outpatient claims in analysis 1, 2, 3. In analysis 4, the outcome will be defined by 1 inpatient or 1 outpatient claims and 1 prescription claim for a symptomatic treatment [donepezil, galantamine, rivastigmine, and memantine] within 6 months of each other with outcome date assigned to second event in the sequence.
- Secondary outcomes: Individual component:

Alzheimer's disease

| Condition | ICD-9 and ICD-10 codes |
|---|---|
| Alzheimer's disease | 331.0*, F00*, G30* |
| Vascular dementia | 290.4*, F01* |
| Senile, presenile, or unspecified dementia | 290.0*, 290.1*. 290.3*, 797*, F03* |
| Dementia in other diseases classified elsewhere | 331.1*, 331.2*, 331.7*, 294.1*, F02* |

For analysis 1,3, and 4 the follow-up will start the day after initiation of <u>Montelukast and Fluticasone</u> and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest
- The date of end of continuous registration in the database,
- End of the study period,

- Measured death event occurs,
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (Montelukast and Fluticasone) plus a defined grace period (i.e., 90 days after the end of the last prescription's days' supply in main analyses).

For analysis 2, the follow-up will start 180 days after initiation of <u>Montelukast and Fluticasone</u> and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- Maximum allowed follow-up time (1095 days) reached

## 7. Propensity score analysis

We will use a propensity-score (PS)¹-based approach to account for measured confounding in this study. The PS will be calculated as the predicted probability of initiating the exposure of interest (i.e., the repurposing candidate) versus the reference drug conditional on baseline covariates using multivariable logistic regression constructed separately in each data source. On average, patients with similar PSs have similar distribution of potential confounders used to estimate the PS. Therefore, analyses conditioned on the PS provide effect estimates that are free from measured confounding. For all our analyses, initiators of each exposure of interest will be matched with initiators of the reference exposure based on their PS within each data source.² Pair matching will be conducted using a nearest-neighbor algorithm, which seeks to minimize the distance between propensity scores in each pair of treated and reference patients,³ and a caliper of 0.025 on the natural scale of the PS will be used to ensure similarity between the matched patients.⁴

We report multiple diagnostics for PS analysis in this protocol. First, the PS distributional overlap is provided between two groups before and after matching to ensure comparability of these groups.<sup>5</sup> Next, balance in each individual covariate between two treatment groups is reported using standardized differences.<sup>6</sup>

# 8. Table for covariate balance

| | Unmatched | | | PS-Matched | | |
|---|---|---|---|---|---|---|
| Variable | Montelukast | Fluticasone | St. Diff | Montelukast | Fluticasone | St. Diff |
| | (N = 12,575) | (N = 38,958) | | (N = 12,572) | (N = 12,572) | |
| Demographics | | | | | | |
| Age, mean (SD) | 72.8 (6.1) | 73.3 (6.4) | -8.20 | 72.8 (6.1) | 72.8 (6.1) | -0.30 |
| Gender, n (%) | | | | | | |
| Male | 3694 (29.4) | 12706 (32.6) | -7.00 | 3694 (29.4) | 3764 (29.9) | -1.20 |
| Female | 8881 (70.6) | 26252 (67.4) | 7.00 | 8878 (70.6) | 8808 (70.1) | 1.20 |
| Race, n (%) | | | | | | |
| White | 10614 (84.4) | 33028 (84.8) | -1.00 | 10613 (84.4) | 10650 (84.7) | -0.80 |
| Black | 831 (6.6) | 3055 (7.8) | -4.80 | 831 (6.6) | 881 (7) | -1.60 |
| Hispanic | 218 (1.7) | 639 (1.6) | 0.70 | 218 (1.7) | 203 (1.6) | 0.90 |
| Other | 912 (7.3) | 2236 (5.7) | 6.10 | 910 (7.2) | 838 (6.7) | 2.30 |
| Region, n (%) | | | | | | |
| Northeast; n (%) | 2271 (18.1) | 8670 (22.3) | ##### | 2271 (18.1) | 2335 (18.6) | -1.30 |
| South; n (%) | 5310 (42.2) | 13528 (34.7) | 15.50 | 5307 (42.2) | 5179 (41.2) | 2.10 |
| Midwest; n (%) | 2498 (19.9) | 8288 (21.3) | -3.50 | 2498 (19.9) | 2546 (20.3) | -1.00 |
| West; n (%) | 2484 (19.8) | 8431 (21.6) | -4.70 | 2484 (19.8) | 2501 (19.9) | -0.30 |
| Other; n (%) | 12 (0.1) | 41 (0.1) | -0.30 | 12 (0.1) | 11 (0.1) | 0.30 |
| Calendar year of index date, n (%) | | | | | | |
| 2014 | 3143 (25) | 10567 (27.1) | -4.90 | 3142 (25) | 3037 (24.2) | 1.90 |
| 2015 | 2585 (20.6) | 8299 (21.3) | -1.80 | 2585 (20.6) | 2519 (20) | 1.30 |
| 2016 | 2396 (19.1) | 7305 (18.8) | 0.80 | 2394 (19) | 2425 (19.3) | -0.60 |
| 2017 | 2330 (18.5) | 6986 (17.9) | 1.50 | 2330 (18.5) | 2408 (19.2) | -1.60 |
| 2018 | 2121 (16.9) | 5801 (14.9) | 5.40 | 2121 (16.9) | 2183 (17.4) | -1.30 |

| Low income subsidy, n (%) | 1824 (14.5) | 6953 (17.8) | -9.10 | 1823 (14.5) | 1859 (14.8) | -0.80 |
|---|---|---|---|---|---|---|
| Dementia risk factors, n (%) | | | | | | |
| Diabetes | 4101 (32.6) | 13257 (34) | -3.00 | 4098 (32.6) | 4087 (32.5) | 0.20 |
| Obesity | 2804 (22.3) | 9138 (23.5) | -2.80 | 2804 (22.3) | 2808 (22.3) | -0.10 |
| Coronary artery disease | 3338 (26.5) | 11429 (29.3) | -6.20 | 3338 (26.6) | 3264 (26) | 1.30 |
| Hypertension | 9870 (78.5) | 30962 (79.5) | -2.40 | 9867 (78.5) | 9909 (78.8) | -0.80 |
| Depression | 2029 (16.1) | 6989 (17.9) | -4.80 | 2029 (16.1) | 2013 (16) | 0.30 |
| Anxiety | 2235 (17.8) | 6921 (17.8) | 0.00 | 2235 (17.8) | 2234 (17.8) | 0.00 |
| Bipolar disorder | 126 (1) | 555 (1.4) | -3.90 | 126 (1) | 120 (1) | 0.50 |
| Schizophrenia | 8 (0.1) | 70 (0.2) | -3.30 | 8 (0.1) | 3 (0) | 1.90 |
| Markers for healthy behavior, frailty, healthcare use | | | | | | |
| Smoking, n (%) | 2803 (22.3) | 10651 (27.3) | ##### | 2803 (22.3) | 2833 (22.5) | -0.60 |
| Mammography, n (%) | 4285 (34.1) | 12152 (31.2) | 6.20 | 4283 (34.1) | 4262 (33.9) | 0.40 |
| Colonoscopy, n (%) | 1465 (11.7) | 4797 (12.3) | -2.00 | 1464 (11.6) | 1465 (11.7) | 0.00 |
| Fecal occult blood test, n (%) | 1172 (9.3) | 3374 (8.7) | 2.30 | 1172 (9.3) | 1172 (9.3) | 0.00 |
| Influenza vaccination, n (%) | 8417 (66.9) | 26819 (68.8) | -4.10 | 8416 (66.9) | 8463 (67.3) | -0.80 |
| Herpes zoster vaccination, n (%) | 3 (0) | 11 (0) | -0.30 | 3 (0) | 2 (0) | 0.60 |
| Pneumococcal vaccination, n (%) | 5584 (44.4) | 17347 (44.5) | -0.20 | 5583 (44.4) | 5680 (45.2) | -1.60 |
| Bone mineral density test, n (%) | 1743 (13.9) | 5139 (13.2) | 2.00 | 1743 (13.9) | 1732 (13.8) | 0.30 |
| Number of distinct prescriptions, mean (SD) | 12.3 (5.8) | 12.5 (5.8) | -2.30 | 12.3 (5.8) | 12.2 (5.7) | 2.00 |
| Number of emergency room visits, mean (SD) | 0.7 (1.4) | 0.8 (1.6) | -8.80 | 0.7 (1.4) | 0.7 (1.2) | 1.20 |
| Number of outpatient visits, mean (SD) | 12.5 (8.4) | 12.4 (8.6) | 1.10 | 12.5 (8.4) | 12.5 (8.6) | 0.90 |
| Number of hospitalizations, mean (SD) | 0.2 (0.6) | 0.2 (0.6) | -6.60 | 0.2 (0.6) | 0.2 (0.5) | 1.40 |

| Number of C-reactive protein tests ordered, mean (SD) | 0.2 (0.8) | 0.2 (0.9) | -1.20 | 0.2 (0.8) | 0.2 (0.8) | 0.40 |
|---|---|---|---|---|---|---|
| Number of serum creatinine tests ordered, mean (SD) | 0.9 (1.6) | 1.1 (2) | ##### | 0.9 (1.6) | 0.9 (1.5) | 1.60 |
| Composite frailty score, mean (SD) | 0.2 (0.1) | 0.2 (0.1) | ##### | 0.2 (0.1) | 0.2 (0.1) | 1.40 |
| Osteoporosis, n (%) | 1911 (15.2) | 5814 (14.9) | 0.80 | 1911 (15.2) | 1912 (15.2) | 0.00 |
| Fractures, n (%) | 877 (7) | 2787 (7.2) | -0.70 | 877 (7) | 893 (7.1) | -0.50 |
| Falls, n (%) | 641 (5.1) | 2326 (6) | -3.80 | 641 (5.1) | 656 (5.2) | -0.50 |
| Use of supplemental oxygen, n (%) | 260 (2.1) | 1091 (2.8) | -4.80 | 260 (2.1) | 279 (2.2) | -1.00 |
| Combined comorbidity score, mean (SD) | 2.2 (2.2) | 2.4 (2.4) | ##### | 2.2 (2.2) | 2.2 (2.2) | 0.50 |
| Comedication use, n (%) | | | | | | |
| Lithium | 17 (0.1) | 50 (0.1) | 0.20 | 17 (0.1) | 12 (0.1) | 1.20 |
| Anti-epileptic mood stabilizers | 142 (1.1) | 562 (1.4) | -2.80 | 142 (1.1) | 149 (1.2) | -0.50 |
| Anti-epileptics (other than mood stabilizers) | 1839 (14.6) | 6087 (15.6) | -2.80 | 1837 (14.6) | 1778 (14.1) | 1.30 |
| Atypical antipsychotics | 170 (1.4) | 719 (1.8) | -3.90 | 170 (1.4) | 158 (1.3) | 0.80 |
| Benzodiazepines | 2537 (20.2) | 7878 (20.2) | -0.10 | 2537 (20.2) | 2523 (20.1) | 0.30 |
| Serotonin-norepinephrine reuptake inhibitors | 715 (5.7) | 2343 (6) | -1.40 | 715 (5.7) | 721 (5.7) | -0.20 |
| Selective serotonin reuptake inhibitors | 2265 (18) | 7367 (18.9) | -2.30 | 2265 (18) | 2205 (17.5) | 1.20 |
| Tricyclic antidepressants (TCAs) | 434 (3.5) | 1548 (4) | -2.80 | 434 (3.5) | 425 (3.4) | 0.40 |
| Typical antipsychotics | 20 (0.2) | 105 (0.3) | -2.40 | 20 (0.2) | 24 (0.2) | -0.80 |
| Anticoagulants | 1163 (9.2) | 4342 (11.1) | -6.30 | 1163 (9.3) | 1217 (9.7) | -1.50 |
| Antiplatelet agents | 947 (7.5) | 3416 (8.8) | -4.50 | 947 (7.5) | 916 (7.3) | 0.90 |
| Nitrates | 915 (7.3) | 3131 (8) | -2.90 | 915 (7.3) | 881 (7) | 1.10 |
| Lipid lowering drugs | 6790 (54) | 22232 (57.1) | -6.20 | 6789 (54) | 6819 (54.2) | -0.50 |
| Non-insulin diabetes medications | 2391 (19) | 7537 (19.3) | -0.80 | 2388 (19) | 2415 (19.2) | -0.50 |

| Insulin | 725 (5.8) | 2740 (7) | -5.20 | 725 (5.8) | 705 (5.6) | 0.70 |
|---|---|---|---|---|---|---|
| Antidepressants | 3634 (28.9) | 11842 (30.4) | -3.30 | 3634 (28.9) | 3557 (28.3) | 1.40 |
| Angiotensin converting enzyme inhibitors (ACEi) | 3269 (26) | 10938 (28.1) | -4.70 | 3268 (26) | 3300 (26.2) | -0.60 |
| Angiotensin II receptor blockers (ARBs) | 3599 (28.6) | 10554 (27.1) | 3.40 | 3598 (28.6) | 3563 (28.3) | 0.60 |
| Beta blockers | 4312 (34.3) | 14499 (37.2) | -6.10 | 4312 (34.3) | 4274 (34) | 0.60 |
| Calcium channel blockers | 3182 (25.3) | 10328 (26.5) | -2.80 | 3181 (25.3) | 3192 (25.4) | -0.20 |
| Disease-modifying antirheumatic drugs (DMARDs) | 457 (3.6) | 1522 (3.9) | -1.40 | 457 (3.6) | 452 (3.6) | 0.20 |
| Diuretics | 5260 (41.8) | 17028 (43.7) | -3.80 | 5259 (41.8) | 5306 (42.2) | -0.80 |
| Biologics (Omalizumab, Mepolizumab,<br>Reslizumab, Benralizumab, Dupilumab) | 89 (0.7) | 218 (0.6) | 1.90 | 89 (0.7) | 77 (0.6) | 1.20 |
| Comorbid conditions, n (%) | | | | | | |
| Atrial fibrillation | 1527 (12.1) | 5492 (14.1) | -5.80 | 1527 (12.1) | 1543 (12.3) | -0.40 |
| Heart failure | 1397 (11.1) | 5145 (13.2) | -6.40 | 1397 (11.1) | 1352 (10.8) | 1.10 |
| Stroke or transient ischemic attack | 858 (6.8) | 3209 (8.2) | -5.40 | 858 (6.8) | 867 (6.9) | -0.30 |
| Peripheral vascular disease | 1056 (8.4) | 3915 (10) | -5.70 | 1055 (8.4) | 1055 (8.4) | 0.00 |
| Hyperlipidemia | 8900 (70.8) | 27637 (70.9) | -0.40 | 8898 (70.8) | 8820 (70.2) | 1.40 |
| Renal dysfunction | 1706 (13.6) | 6279 (16.1) | -7.20 | 1705 (13.6) | 1704 (13.6) | 0.00 |
| Chronic liver disease | 810 (6.4) | 2628 (6.7) | -1.20 | 809 (6.4) | 807 (6.4) | 0.10 |
| Ischemic heart disease | 3250 (25.8) | 11107 (28.5) | -6.00 | 3250 (25.9) | 3170 (25.2) | 1.50 |
| Chronic obstructive pulmonary disease | 5222 (41.5) | 16890 (43.4) | -3.70 | 5220 (41.5) | 5213 (41.5) | 0.10 |
| Malignancy | 3369 (26.8) | 11073 (28.4) | -3.70 | 3369 (26.8) | 3411 (27.1) | -0.80 |
| Drug or alcohol abuse or dependence | 944 (7.5) | 4336 (11.1) | ##### | 944 (7.5) | 936 (7.4) | 0.20 |
| Venous thromboembolism | 425 (3.4) | 1565 (4) | -3.40 | 425 (3.4) | 423 (3.4) | 0.10 |
| Rheumatoid Arthritis | 595 (4.7) | 1994 (5.1) | -1.80 | 595 (4.7) | 592 (4.7) | 0.10 |

| Other Asthma treatments and Asthma | | | | | | |
|---|---|---|---|---|---|---|
| severity indicators Asthma exacerbation, n (%) | 213 (1.7) | 478 (1.2) | 3.90 | 211 (1.7) | 174 (1.4) | 2.40 |
| Bronchiectasis, n (%) | 347 (2.8) | 1006 (2.6) | 1.10 | 346 (2.8) | 357 (2.8) | -0.50 |
| Interstitial lung disease, lung fibrosis, ARDS, n (%) | 1220 (9.7) | 3941 (10.1) | -1.40 | 1219 (9.7) | 1205 (9.6) | 0.40 |
| Lung Cancer, n (%) | 144 (1.1) | 674 (1.7) | -4.90 | 144 (1.1) | 137 (1.1) | 0.50 |
| Pneumonia, n (%) | 694 (5.5) | 2455 (6.3) | -3.30 | 693 (5.5) | 670 (5.3) | 0.80 |
| Pulmonary Hypertension, n (%) | 194 (1.5) | 691 (1.8) | -1.80 | 194 (1.5) | 182 (1.4) | 0.80 |
| Respiratory failure, n (%) | 723 (5.7) | 2725 (7) | -5.10 | 722 (5.7) | 704 (5.6) | 0.60 |
| Sarcoidosis, n (%) | 60 (0.5) | 259 (0.7) | -2.50 | 60 (0.5) | 68 (0.5) | -0.90 |
| Tuberculosis, n (%) | 2157 (17.2) | 7552 (19.4) | -5.80 | 2155 (17.1) | 2177 (17.3) | -0.50 |
| Acute Upper/ Lower Respiratory Tract infection, n (%) | 4789 (38.1) | 14315 (36.7) | 2.80 | 4788 (38.1) | 4850 (38.6) | -1.00 |
| Pulmonary function test, n (%) | 4989 (39.7) | 13566 (34.8) | 10.00 | 4988 (39.7) | 4943 (39.3) | 0.70 |
| Number of Pulmonologist visits, mean (SD) | 1.1 (2.4) | 1 (2.5) | 3.50 | 1.1 (2.4) | 1.1 (2.5) | 0.90 |
| Antibiotics, n (%) | 9638 (76.6) | 29724 (76.3) | 0.80 | 9636 (76.6) | 9601 (76.4) | 0.70 |
| Corticosteroids, n (%) | 6750 (53.7) | 18540 (47.6) | 12.20 | 6748 (53.7) | 6551 (52.1) | 3.10 |
| ICS (excluding Fluticasone), n (%) | 3647 (29) | 8369 (21.5) | 17.40 | 3644 (29) | 3386 (26.9) | 4.60 |
| LAMA, n (%) | 884 (7) | 3315 (8.5) | -5.50 | 884 (7) | 883 (7) | 0.00 |
| LABA, n (%) | 2532 (20.1) | 12953 (33.2) | ##### | 2532 (20.1) | 2143 (17) | 8.00 |
| Leukotriene receptor antagonist (excluding Montelukast), n (%) | 93 (0.7) | 150 (0.4) | 4.70 | 91 (0.7) | 68 (0.5) | 2.30 |
| SABA, n (%) | 6687 (53.2) | 21764 (55.9) | -5.40 | 6684 (53.2) | 6657 (53) | 0.40 |
| SAMA, n (%) | 656 (5.2) | 2193 (5.6) | -1.80 | 656 (5.2) | 629 (5) | 1.00 |

## 9. Statistical analysis plans

Incidence rates for the outcome will be estimated for the treatment and reference groups before and after PS matching. The competing risk of death could be of concern for the current set of analyses if mortality is frequent among patients included in the cohort and if differences in the risk of mortality between treatment and reference groups are substantial. In the PS-matched sample, we will use cause-specific hazard models<sup>7</sup> to provide hazard ratios averaged over the entire follow-up period as well as interval specific hazard ratios (1, 2, and 3 years) for the association between the treatment of interest and risk of ADRD after considering all-cause mortality as a competing event. Pre-specified subgroup analyses will be conducted based on age, sex, and baseline cardiovascular disease.

## 10. References

- **1.** Rosenbaum PR, Rubin DB. The central role of the propensity score in observational studies for causal effects. *Biometrika*. 1983;70(1):41-55.
- 2. Rassen JA, Avorn J, Schneeweiss S. Multivariate-adjusted pharmacoepidemiologic analyses of confidential information pooled from multiple health care utilization databases. *Pharmacoepidemiology and drug safety.* 2010;19(8):848-857.
- **3.** Rassen JA, Shelat AA, Myers J, Glynn RJ, Rothman KJ, Schneeweiss S. One-to-many propensity score matching in cohort studies. *Pharmacoepidemiol Drug Saf.* May 2012;21 Suppl 2:69-80.
- **4.** Austin PC. Some Methods of Propensity-Score Matching had Superior Performance to Others: Results of an Empirical Investigation and Monte Carlo simulations. *Biometrical Journal*. 2009;51(1):171-184.
- **5.** AM Walker AM, Patrick A, Lauer M, et al. Tool for Assessing the Feasibility of Comparative Effectiveness Research. *Comp Effect Res* 2013;3:11-20.
- **6.** Franklin JM, Rassen JA, Ackermann D, Bartels DB, Schneeweiss S. Metrics for covariate balance in cohort studies of causal effects. *Statistics in medicine*. May 10 2014;33(10):1685-1699.
- **7.** Austin PC, Lee DS, Fine JP. Introduction to the analysis of survival data in the presence of competing risks. *Circulation*. 2016;133(6):601-609.